CLINICAL TRIAL: NCT03595514
Title: A Randomized Comparison Between Single- and Double-injection Ultrasound-Guided Costoclavicular Block
Brief Title: Single Versus Double Injection Costoclavicular Block
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Collaborators: University of Chile (Other)
Responsible Party: Principal Investigator, De Tran, Professor, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: MUHC 2019-4673
Record Dates: First submitted 2018-07-01; First posted 2018-07-23 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Upper Extremity Injury
MeSH Terms: conditions — Arm Injuries | interventions — Injections; Lidocaine; Bupivacaine; Epinephrine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Randomized
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants will not be allowed to see the ultrasound screen. Outcome assessors will not be present during the performance of the block.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Injection (Active Comparator): Local anesthetic injection with a mixture of 35 mL of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL and dexamethasone 2 mg, in the middle of the three cords of the brachial plexus
  Interventions: Other: Single injection; Drug: lidocaine, bupivacaine, epinephrine, dexamethasone
- Double Injection (Experimental): Local anesthetic injection with a mixture of 35 mL of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL and dexamethasone 2 mg, in the middle of the three cords of the brachial plexus as well as at the intersection of the subclavian artery and the medial cord.
  Interventions: Other: Double injection; Drug: lidocaine, bupivacaine, epinephrine, dexamethasone

INTERVENTIONS:
Other: Single injection — Local anesthetic injection with a mixture of 35 mL of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL and dexamethasone 2 mg, in the middle of the three cords of the brachial plexus
  Arms: Single Injection
Other: Double injection — Local anesthetic injection with a mixture of 35 mL of lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL and dexamethasone 2 mg, in the middle of the three cords of the brachial plexus as well as at the intersection of the subclavian artery and the medial cord.
  Arms: Double Injection
Drug: lidocaine, bupivacaine, epinephrine, dexamethasone — lidocaine 1.0%-bupivacaine 0.25% with epinephrine 5 µ/mL and dexamethasone

SUMMARY:
In this trial, the objective is to compare single- and double-injection ultrasound-guided costoclavicular blocks. The rationale behind this idea is that a second local anesthetic injection, inside the costoclavicular space, may compensate for the dynamic cord dispersion seen with the single-injection technique. Thus the research hypothesis is that, compared to its single-injection counterpart, a double injection costoclavicular block will result in a shorter onset time.

DETAILED DESCRIPTION:
The costoclavicular block (CCB) constitutes a relatively novel technique for infraclavicular brachial plexus blockade, whereby local anesthetics (LAs) are injected inside the costoclavicular space. In this location, the 3 cords of the brachial plexus are very tightly clustered together; this topography would theoretically result in a very swift brachial plexus block Unfortunately, in two recent trials comparing CCB and conventional infraclavicular brachial plexus block, the authors were unable to detect differences in success rate, onset times and LA requirement between the 2 methods. It could be speculated that the explanation resides in dynamic cord dispersion. With CCB, the initial needle target lies in the middle of the 3 cords of the brachial plexus. However, with LA injection, the cords can quickly migrate away from each other. Thus, the anatomical benefits conveyed by the initial compact topography may be lost.

In this trial, the objective is to compare single- and double-injection ultrasound-guided costoclavicular blocks. The rationale behind this idea is that a second local anesthetic injection, inside the costoclavicular space, may compensate for the dynamic cord dispersion seen with the single-injection technique. Thus the research hypothesis is that, compared to its single-injection counterpart, a double injection costoclavicular block will result in a shorter onset time.

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 75 years
* American Society of Anesthesiologists classification 1-3
* body mass index between 18 and 30

Exclusion Criteria:

* adults who are unable to give their own consent
* pre-existing neuropathy (assessed by history and physical examination)
* coagulopathy (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. platelets ≤ 100, International Normalized Ratio ≥ 1.4 or partial thromboplastin time ≥ 50)
* renal failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. creatinine ≥ 100)
* hepatic failure (assessed by history and physical examination and, if deemed clinically necessary, by blood work up i.e. transaminases ≥ 100)
* allergy to local anesthetic
* pregnancy
* prior surgery in the infraclavicular costoclavicular region
* chronic pain syndromes requiring opioid intake at home

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2018-07-30 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Onset time of brachial plexus blockade | Within 30 minutes of block performance
  Onset until a minimal composite score of 14 points in a scale of 0-16 points, evaluating sensitive and motor function of each 4 terminal branches.

SECONDARY OUTCOMES:
Performance time during the brachial plexus block | Intraoperative (During block performance)
  the sum of: 1. the acquisition time of the sonographic image and 2. the time to perform block itself (from skin anesthesia to the end of LA injection)
Number of needle passes | Intraoperative (During block performance)
  The initial needle insertion counted as the first pass. Any subsequent needle advancement that is preceded by a retraction of at least 10 mm counts as an additional pass
Procedure pain during the brachial plexus block | Intraoperative (During block performance)
  Pain reported during procedure, rated acording to a visual rating scale from 0 to 10 points (0= no pain and 10= worst imaginable pain)
Incidence of surgical anesthesia | Thirty minutes after block performance
  Incidence of surgeries performed without the supplemental use of local anesthetics infiltration, narcotics or general anesthesia
Incidence of Adverse events | Intraoperative (During block performance)
  Incidence of adverse events related to brachial plexus block ((paresthesia, vascular puncture, hematoma, Horner syndrome, pneumothorax)

CONTACTS AND LOCATIONS:
Overall Officials: De Q Tran, MD, FRCPC, Principal Investigator — McGill University Health Centre/Research Institute of the McGill University Health Centre
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Layera S, Aliste J, Bravo D, Fernandez D, Garcia A, Finlayson RJ, Tran DQ. Single- versus double-injection costoclavicular block: a randomized comparison. Reg Anesth Pain Med. 2020 Mar;45(3):209-213. doi: 10.1136/rapm-2019-101167. Epub 2020 Jan 14. PMID 31941792